CLINICAL TRIAL: NCT02128880
Title: A Randomized Clinical Trial of the Contraception and Alcohol Risk Reduction Internet Intervention to Reduce AEP Risk in Community Women
Brief Title: Contraception and Alcohol Risk Reduction Internet Intervention Randomized Trial
Acronym: CARRII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, Associate Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17319; R34AA020853 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: AEP, drinking, contraception, FASD, Internet interventions
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARRII (Experimental): CARRII: This is a highly interactive Internet intervention consisting of 6 Cores of Intervention material, including Core 1, Overview, Core 2: Your Risk for AEP, Core 3: Drinking, Core 4: Contraception, Core 5: Thoughts and Decisions, and Core 6: Commit to It.
  Interventions: Behavioral: CARRII
- Patient Education (Active Comparator): CARRII Education: This is a static website containing educational information on the following topics: What is Alcohol Exposed Pregnancy (AEP)?, Fetal Alcohol Spectrum Disorders, Impact of AEP, Prevalence of AEP, Causes and Prevention of AEP, Treatment for AEP, and Links to related information.
  Interventions: Behavioral: CARRII Education

INTERVENTIONS:
Behavioral: CARRII — CARRII is an interactive, personalized and tailored Internet intervention designed to reduce the risk of AEP among drinking women of childbearing age.
  Arms: CARRII
Behavioral: CARRII Education — CARRII Education provides information on women's health related to drinking and contraception in a static website format.
  Other Names: Patient Ed
  Arms: Patient Education

SUMMARY:
The goal of the proposed research is to develop and pilot test a novel Internet intervention to reduce the risk of Alcohol-exposed pregnancy (AEP). Efficacious interventions to reduce the risk of AEP have been developed, but are not widely available. In this project, we will develop a novel Internet intervention to reduce AEP risk by combining the resources of two research teams focused on primary prevention of Fetal Alcohol Spectrum Disorders (FASD) and robust Internet interventions, respectively. We will use our evidence-based AEP risk reduction intervention materials and our existing Internet intervention development platform to build and pilot test an Internet intervention (Contraception and Alcohol Risk Reduction Internet Intervention, CARRIII) in a stage 1 behavioral and integrative therapies development project.

This three year R34 project will develop and program the new Internet intervention, and will determine the feasibility and preliminary efficacy of the intervention in a pilot RCT. In this protocol, we will assess the feasibility and preliminary efficacy of CARRIII against a Patient Education Website condition in a pilot randomized clinical trial (RCT) with assessments at pre-, post-, and 6 months.The primary hypothesis is that women randomized to the CARRIII condition will change more in 3 markers of AEP-related outcomes (risky drinking, ineffective contraception, and AEP risk) than women assigned to the Patient Education website condition. We will prepare for a future cost effectiveness evaluation in the larger RCT to follow by pilot testing proposed measures. The pilot RCT will yield effect size estimates for a subsequent fully powered trial. If the Internet intervention is promising, it should be tested in a fully powered national trial. The Internet intervention could substantially increase the options for AEP prevention, and could lead to a reduction in incident FASD.

DETAILED DESCRIPTION:
As the first study of a fully interactive Internet intervention for reducing AEP risk, the proposed project is a significant extension of the growing literature on Internet interventions to reduce problem drinking, which established their feasibility and acceptability, with evidence of efficacy especially in the university drinking setting. Most brief online interventions for problem drinking have incorporated self-assessment and tailored normative feedback, and some offer cognitive behavioral exercises. Only one web-based intervention to date targeted AEP risk. In that study, a static Internet presentation of AEP risk reduction intervention materials was compared to the same intervention delivered by mail in a quasi-experimental design. The web delivered and mailed versions of this self-guided change intervention significantly reduced AEP risk. The proposed intervention will build on this study as well as existing alcohol Internet intervention findings and extend the focus to a new population with a new goal (AEP prevention) by targeting both drinking AND ineffective contraception. It will also incorporate significant enhancements compared to the static web-based self-guided change intervention for AEP by adding dynamic, interactive, and feedback elements that mirror the interaction in successful face-to-face interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-44 who are fertile

  * can provide informed consent
  * are at risk for unintended pregnancy due to ineffective, inconsistent, or absent contraception in the past 3 months
  * speak and read English
  * have more than 1 episode of drinking 4 or more standard drinks/day during the past 3 months
  * have regular access to a computer, the Internet, and telephone
  * reside in the US.

Exclusion Criteria:

* • Currently pregnant or planning pregnancy in the next 6 months

  * cognitive disorders including mental retardation and dementia that could impair ability to understand the intervention material or give informed consent, or psychotic disorder due to the same issues
  * live outside the US

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Drinks per drinking day (DDD) | 90 day
  The primary outcome will be drinks per drinking day measured by the combination of prospective self-report diaries and the Time-Line Follow-Back (TLFB) 90 day retrospective self-report, with a secondary outcome of episodes of ineffective contraception.

SECONDARY OUTCOMES:
Ineffective contraception rate | 90 day
  The primary outcome will be drinks per drinking day measured by the combination of prospective self-report diaries and the Time-Line Follow-Back (TLFB) 90 day retrospective self-report, with a secondary outcome of episodes of ineffective contraception.

OTHER OUTCOMES:
Alcohol-exposed pregnancy risk | 90-day
  This variable is determined by the combination of drinking risk and pregnancy risk.

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Ingersoll, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- Behavioral Health and Technology Lab, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Behavioral Health and Technology Lab at University of Virginia — http://bht.virginia.edu/